CLINICAL TRIAL: NCT07374302
Title: REAPPRAISED: Riociguat in Triple Therapy for Pulmonary Arterial Hypertension - A Single-Center Retrospective Study With Composite Endpoint Evaluation
Brief Title: Riociguat in Triple Therapy for Pulmonary Arterial Hypertension in Real-World Practice
Acronym: REAPPRAISED
Status: Not yet recruiting | Type: Observational
Sponsor: Caio Júlio César dos Santos Fernandes (Other)
Responsible Party: Sponsor-Investigator, Caio Júlio César dos Santos Fernandes, Principal investigator, University of Sao Paulo General Hospital
Organization: University of Sao Paulo General Hospital (Other)
Other Study IDs: SGP 27906
Record Dates: First submitted 2026-01-12; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary Arterial Hypertension; Riociguat; Triple Therapy; Real-World Evidence; PDE5 Inhibitor Switch; Observational Study
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Riociguat Triple Therapy Cohort: Adult patients with pulmonary arterial hypertension receiving triple therapy who switched from a phosphodiesterase-5 inhibitor to riociguat as part of routine clinical care. The index date (T0) is defined as the date of riociguat initiation.

SUMMARY:
Pulmonary arterial hypertension is a rare and serious disease that can lead to heart failure and early death despite modern treatments. Many patients are treated with a combination of medications targeting different disease pathways, but some continue to have an inadequate response.

Riociguat is a medication that acts on the nitric oxide pathway and may be beneficial in patients who do not respond well to phosphodiesterase-5 inhibitors. In routine clinical practice, some patients receiving triple therapy switch from a phosphodiesterase-5 inhibitor to riociguat.

The REAPPRAISED study evaluates outcomes in patients with pulmonary arterial hypertension who switched to riociguat while receiving triple therapy. This observational study uses data from routine clinical care and does not involve any experimental treatment. The results may help improve understanding of the effectiveness and safety of this treatment strategy in real-world practice.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH) is a progressive disease associated with high morbidity and mortality despite the use of combination therapy. Triple therapy including an endothelin receptor antagonist, a prostacyclin pathway agent, and a phosphodiesterase-5 inhibitor is commonly used; however, a subset of patients shows an inadequate clinical response.

Riociguat is a soluble guanylate cyclase stimulator that increases cyclic GMP through both nitric oxide-dependent and nitric oxide-independent mechanisms. Switching from a phosphodiesterase-5 inhibitor to riociguat has shown clinical benefit in selected patients, but data in real-world settings and in patients already receiving triple therapy remain limited.

REAPPRAISED is a single-center, retrospective, observational study conducted in a pulmonary hypertension referral center. The study evaluates clinical outcomes following the switch from a phosphodiesterase-5 inhibitor to riociguat in patients with PAH receiving triple therapy. All treatment decisions were made by the treating physicians as part of routine clinical care. No study-mandated interventions or treatment assignments were performed, and data were obtained from medical records.

ELIGIBILITY:
Inclusion Criteria

* Adults aged 18 years or older.
* Confirmed diagnosis of pulmonary arterial hypertension (Group 1).
* Treatment with triple therapy including an endothelin receptor antagonist, a prostacyclin pathway agent, and a phosphodiesterase-5 inhibitor for at least 12 weeks.
* Switch from a phosphodiesterase-5 inhibitor to riociguat as part of routine clinical care.
* Availability of minimum data to assess the primary outcome at 6 months.

Exclusion Criteria

* Concomitant use of phosphodiesterase-5 inhibitors and riociguat.
* Inability to confirm vital status or hospitalization outcomes within 6 months.
* Participation in an interventional clinical trial that mandated the treatment switch.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adult patients with pulmonary arterial hypertension receiving triple therapy who switched from a phosphodiesterase-5 inhibitor to riociguat in routine clinical practice at a specialized referral center. All patients were followed using retrospective data from medical records to assess clinical outcomes, safety, and treatment persistence. No study-related interventions were performed.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite Clinical Outcome at 6 Months | 6 months (24±8 weeks) after switch
  Composite clinical outcome assessed at 6 months (24±8 weeks) after the switch to riociguat, defined as achievement of at least two of the following criteria: improvement in six-minute walk distance of at least 10% or 30 meters; World Health Organization functional class I or II; and reduction in BNP levels of at least 30%, in the absence of clinical worsening. Clinical worsening is defined as all-cause mortality, hospitalization due to pulmonary arterial hypertension, or unplanned therapeutic escalation.

SECONDARY OUTCOMES:
Persistence and Time to Discontinuation of Riociguat | Up to 6 months
  reatment persistence at 6 months and time to discontinuation of riociguat for any reason.
Safety Outcomes | Up to 6 months
  Occurrence of adverse events, including symptomatic hypotension, syncope, serious adverse events, and treatment interruptions due to adverse events.
Health Care Utilization | 6 months before and 6 months after switch
  Occurrence of hospitalizations due to pulmonary arterial hypertension and emergency visits in the 6 months before and after the switch to riociguat.
Functional Changes | From baseline to 6 months
  Changes in functional level before and after the switch to riociguat.
Risk Stratification (COMPERA 2.0) | From baseline to 6 months
  Changes in risk stratification using the COMPERA 2.0 score, when sufficient data are available.

CONTACTS AND LOCATIONS:
Overall Officials: Caio Fernandes, MD, Principal Investigator — UNIVERSIDADE SAO PAULO

IPD SHARING:
Plan to Share IPD: No